CLINICAL TRIAL: NCT03833076
Title: Evaluation of Performance and Safety of a New Medical Device Class IIb Not Yet CE Marked in Proctological Disorders: a Randomised, Double-blind, Parallel-groups, Multicentric, Placebo-controlled, Prospective Clinical Study.
Brief Title: A New Class IIb MD in Proctological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathura S.p.A (Industry)
Collaborators: Evidilya S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ProctoMD01
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Proctological Disorders

STUDY DESIGN:
Intervention Model Description: a randomised, double-blind, parallel-groups, multicentric, placebo-controlled, prospective clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A: Medical Device Procto (Experimental): Medical device Procto presents itself as a translucent green gel with a typical smell; it is intended for topical use.
  Posology: external or internal use by means of the provided rectal applicator and following the instructions on the package insert. It can be applied when needed, after intimate cleansing, at any time.
  Interventions: Device: Medical device Procto
- GROUP B: Matching placebo (Placebo Comparator): Investigational Product (IP) placebo presents itself as a translucent green gel with a typical smell; it is intended for topical use.
  Posology: external or internal use by means of the provided rectal applicator and following the instructions on the package insert. It can be applied when needed, after intimate cleansing, at any time.
  Interventions: Device: Matching placebo

INTERVENTIONS:
Device: Medical device Procto — Medical device Procto presents itself as a translucent green gel with a typical smell.
  Arms: GROUP A: Medical Device Procto
Device: Matching placebo — IP placebo presents itself as a translucent green gel with a typical smell.
  Arms: GROUP B: Matching placebo

SUMMARY:
The aim of this study is primarily to investigate the performance of a new medical device not yet CE marked in comparison with placebo, in relieving proctological symptomatology in adult patients reporting symptoms of hemorrhoids (grade 1-3), anal fissures and proctitides.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged between 18 and 75 years.
2. Patients reporting symptoms of haemorrhoids (grade 1-3*), anal fissures and proctitides or already diagnosed with haemorrhoids (grade 1-3), anal fissures and proctitides; diagnosis confirmed by proctological examination at Screening Visit.

   *Grade 1 - Haemorrhoid protrudes into the anal canal but does not prolapse outside the anus.

   Grade 2 - Haemorrhoid protrudes through the anus during straining or evacuation but returns spontaneously.

   Grade 3 - Haemorrhoid protrudes through the anus during straining or evacuation but needs to be manually returned to position.

   Grade 4 - Haemorrhoid remains prolapsed outside of the anus.
3. Patients agreeing not to use any other systemic or topic medicinal / product to treat haemorrhoids, anal fissures and proctitides during the study and not to modify their personal hygiene products.
4. Female patients of childbearing potential following a reliable contraceptive method (according to Investigator's opinion).
5. Willingness to participate in the study and to sign an informed consent form.

Exclusion Criteria:

1. Patients presenting infective anal or rectal pathologies (in particular bacterial infections associated with proctitides or proctitides caused by viral infections).
2. Patients presenting complicated haemorrhoids.
3. Patients with Crohn's disease or malignancy.
4. Patients presenting undiagnosed abnormal rectal bleeding.
5. Patients with known or suspected rectal hypersensitivity.
6. Patients presenting coagulation disorders or on anticoagulant drug therapy (except clopidogrel or acetylsalicylic acid).
7. Patients in treatment with topic or systemic medications / products to treat haemorrhoids, fissures and proctitides, currently or in the 2 weeks prior to Screening Visit.
8. Patients using laxatives or stool softener currently or in the 2 weeks prior to Screening Visit.
9. Patients pregnant or breastfeeding.
10. Patients reporting past or present narcotic addiction or alcoholism.
11. Patients that participated in any other clinical trial during the last month or participating in any clinical trial while participating in this trial.
12. Patients reporting allergy or intolerance to any component of test product, placebo or rescue product.
13. Patients who in the opinion of the principal Investigator are at risk of non-compliance to the study procedures or who are otherwise not appropriate to include in this clinical trial.
14. Patients presenting contraindications to Proktis-M (rescue product), according to concerning leaflet.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Assessment of symptoms according to the Proctological Symptom Scale (PSS) | from Day 0 to Day 14
  Assessment of symptoms according to the Proctological Symptom Scale - PSS (according to 100 mm Visual Analogue Scales; from "no symptoms" to "overwhelming symptoms); comparison between groups, from Day 0 to Day 14

SECONDARY OUTCOMES:
Investigator's assessment of signs | from Day 0 to Day 14
  Investigator's assessment of signs: anal pain, inflammation and visible bleeding, categorized as none, mild, moderate, or severe (corresponding to a score of 0, 1, 2 or 3, respectively); comparison between groups, from Day 0 to Day 14.
Assessments done by Investigator of overall improvement | from Day 0 to Day 14
  Assessments done by Investigator of overall improvement by means of Global Assessment of Improvement (GAI - according to a 7-grade scoring system, 0-6); comparison between groups, at Day 14.
Self-assessment of subjective symptoms | from Day 0 to Day 14
  Self-assessment of subjective symptoms (anal pain, pain or discomfort during evacuation, itching, irritation or inflammation, bleeding) by means of 100 mm Visual Analogue Scales (from "no symptoms" to "overwhelming symptoms"); comparison between groups, from Day 0 to Day 14.
Self-assessment of overall treatment | from Day 0 to Day 14
  Self-assessment of overall treatment by means of Overall Treatment Evaluation (OTE - according to a 15-point scale; from -7 to -1 = worse; 0 = no change; from +1 to +7 = better); comparison between groups, at Day 14.
Patient willingness | from Day 0 to Day 14
  Patient willingness to use the product in the future, assessed on 1 - 4 points scale (strongly disagree=1, disagree=2, agree=3, strongly agree=4); comparison between groups, at Day 14.
Assessment of rescue product | from Day 0 to Day 14
  Assessment of rescue product use (starting date the rescue product was used); comparison among groups, at Day 14.
Assessment of rescue product | from Day 0 to Day 14
  Assessment of rescue product use (number of times the rescue product was used); comparison among groups, at Day 14.

CONTACTS AND LOCATIONS:
Locations (1):
- Isituto Clinico Humanitas, Rozzano, Milano, Italy